CLINICAL TRIAL: NCT02089412
Title: A Study to Determine the Effect of a High-Fat Meal on the Rate and Extent of E2006 Absorption in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2006-A001-008
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Subjects
Keywords: Healthy Subjects; Absorption; High-Fat Meal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E2006: fed conditions (Experimental): E2006 10-mg will be administered as a single dose under fed treatment conditions.
  Interventions: Drug: E2006
- E2006: fasted conditions (Experimental): E2006 10-mg will be administered as a single dose under fasted treatment conditions.
  Interventions: Drug: E2006

INTERVENTIONS:
Drug: E2006

SUMMARY:
This is an open-label, single-dose, randomized crossover study of single oral 10-mg tablet doses administered either after an overnight fast or in combination with a standard high-fat meal in healthy subjects.

DETAILED DESCRIPTION:
The study will have 2 phases: Prerandomization and Randomization. The Prerandomization Phase will consist of 2 periods: Screening and Baseline (Baseline Period 1), during which each subject�s study eligibility will be determined and baseline assessments will be conducted. During this phase, each eligible subject will be randomized to 1 of 2 treatment sequences to receive single oral doses of E2006 10 mg under fasted and fed conditions. The Randomization Phase will consist of 3 periods: administration of the first randomized dose (Treatment Period 1), baseline for the second randomized dose (Baseline Period 2), and administration of the second randomized dose (Treatment Period 2).

ELIGIBILITY:
Inclusion Criteria

1. Healthy males or females, ages 18 to 55 years
2. Body mass index greater than 18 and less than or equal to 32 kg/m2 at Screening
3. All females must be of nonchildbearing potential, defined as postmenopausal women (defined as at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause) or subjects who have been sterilized surgically or who are otherwise proven sterile (eg, bilateral tubal ligation with surgery at least 6 months prior to dosing, hysterectomy, or bilateral oophorectomy with surgery at least 2 months prior to dosing). In addition, females must have a negative serum B-human chorionic gonadotropin test result at Screening.
4. Males who are not abstinent or have undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use a highly effective method of contraception (eg, condom plus spermicide, condom plus diaphragm with spermicide, intrauterine device starting at least 1 menstrual cycle prior to starting study drug and throughout the entire study period and for 30 days [longer if appropriate] after the last dose of study drug)
5. Are willing and able to comply with all aspects of the protocol
6. Provide written informed consent

Exclusion Criteria

1. Any subject that has a known history of malaria or has traveled to a country with known malarial risk (ie, is designated as "high" or "moderate" risk country according to the list available at http://www.cdc.gov/malaria) within the last year
2. Subjects with a history of bowel resection, any malabsorptive disorder, severe gastroparesis, or any gastrointestinal procedure for the purpose of weight loss (including Lapband(TM)), which would slow gastric emptying and potentially affect PK profiles of E2006
3. Subjects with a known history of clinically significant drug or food allergies or a known allergy or hypersensitivity to capsule or tablet ingredients
4. Subjects who experienced a weight loss or gain of greater than 10% between Screening and prior to dosing
5. Subjects who had a clinically significant illness that required medical treatment within 8 weeks or a clinically significant infection within 4 weeks of dosing
6. Subjects with any clinically abnormal symptom or organ impairment found in medical history, symptoms or signs, vital sign measurements, electrocardiogram (ECG) findings, or laboratory test results that require medical treatment found in medical history or at screening and baseline
7. Subjects known to be positive for human immunodeficiency virus, or subjects who have positive hepatitis B or hepatitis C screening test results
8. Subjects who have a history of drug or alcohol dependency or abuse (as defined by The Diagnostic and Statistical Manual of Mental Disorders V criteria) within approximately 2 years prior to Screening, or who have a positive urine drug test result at Screening or Baseline
9. Subjects who received blood products within 4 weeks, donated blood within 8 weeks, or donated plasma within 1 week of dosing
10. Subjects who used hormonal replacement therapy within 3 months prior to dosing
11. Subjects who used any drugs, over-the-counter medications, nutritional supplements (eg, products containing St. John's wort), excessive doses of vitamins (in the opinion of the principal investigator), herbal preparations, or foods or beverages known to modulate cytochrome P450 ([CYP] eg, CYP3A4) or transporters within 4 weeks prior to dosing, or who are unwilling to abstain from using these during the study
12. Subjects who engaged in intense physical activity within 1 week prior to Baseline (eg, weight training)
13. Subjects who smoke or have used tobacco- or nicotine-containing products within 3 months prior to dosing
14. Subjects who habitually consume more than 400-mg caffeine per day
15. Subjects who participated (received investigational product) in another clinical trial less than 1 month (or 5 elimination half-lives of the investigational product) prior to dosing or who are currently enrolled in another clinical trial
16. Subjects with a disease that may influence the outcome of the study, such as psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism, or subjects who have any condition that would make him or her, in the opinion of the investigator, unsuitable for the study or who, in the opinion of the investigator, are not likely to complete the study for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of E2006: AUC(t-0) | Up to Day 15 (336 hours)
Pharmacokinetics of E2006: AUC(t-inf) | Up to Day 15 (336 hours)
Pharmacokinetics of E2006: Maximum Concentration (Cmax) | Up to Day 15 (336 hours)
Pharmacokinetics of E2006: time attain to Cmax (tmax) | Up to Day 15 (336 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development LLC, Austin, Texas, United States